CLINICAL TRIAL: NCT05050201
Title: Implementation of a Digital Cognitive Behavioural Therapy Intervention for Insomnia in First Episode Psychosis in the Context of Covid19: A Mixed Methods Study
Brief Title: Implementation of Digital CBT for Insomnia in First Episode Psychosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other); Big Health Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GN21MH015
Record Dates: First submitted 2021-08-05; First posted 2021-09-20 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Insomnia; Psychosis; First Episode Psychosis
Keywords: insomnia; psychosis; first episode psychosis; digital CBT; CBT-I
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: All service users who would like to trial the Sleepio intervention will be able to do so.
Masking Description: Participation is not masked - any service users who would like to participate may do so and their keyworker will be notified as a mandatory condition of consent
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sleepio Intervention (Experimental): Participants using the Sleepio application - access for 6 sessions, over 10 weeks
  Interventions: Device: Sleepio

INTERVENTIONS:
Device: Sleepio — Digital CBT application for insomnia

SUMMARY:
This study uses mixed methods to investigate the implementation of digital cognitive behavioural therapy for insomnia (Sleepio) in a first episode of psychosis service (FEP). Interviews will be conducted with keyworker clinicians and service users to consider their expectations for digital sleep intervention. The rates of recruitment into the study, eligibility, completion of baseline measures, completion of the intervention sessions, attrition from the intervention and completion of follow up measures will be recorded. Interviews will be conducted with keyworker clinicians and service users to consider their experiences of digital sleep intervention.

The primary outcome will be a logic model describing factors acting upon the implementation of Sleepio in this population. The investigators will provide signal data in relation to changes in insomnia severity, psychosis symptomatology, and general mental health.

DETAILED DESCRIPTION:
First episode psychosis (FEP) services present a unique opportunity to effect change in outcomes in those affected by experiences of psychosis. Sleep disorder, particularly insomnia, is common in those affected by psychosis, including those experiencing a first episode and are associated with increased symptomatology. Mood and worry mediate the relationship between sleep and psychosis symptomatology and research suggests that improving sleep in this population can improve mental health symptomatology and longer term outcomes. Cognitive Behavioural Therapy is effective in treating insomnia (CBT-I). Pilot research suggests that insomnia is a tractable clinical target in psychosis. Furthermore, there is an appetite for therapeutic interventions for sleep in this population.

"Sleepio" is an online Cognitive Behavioural Therapy for Insomnia (CBT-I) programme. Sleepio's components are those common to CBT-I interventions: i) Psychoeducation on sleep hygiene and processes; ii) cognitive components including restructuring, mindfulness, positive imagery, paradoxical intention training (trying to stay awake), and resolving thoughts about one's day; and iii) behavioural components including sleep restriction, stimulus control, and relaxation techniques. Sleepio is composed of six 20-minute sessions presented by an animated therapist ("the Professor"), which are unlocked weekly. Participants complete an initial assessment (please see 'Sleepio Onboarding Questions') and chose a treatment goal, which drives initial personalisation of the application. Participants book digital 'appointments' with the Professor and receive prompts to complete these 6 sessions, to enter sleep data and to complete the Sleep Condition Indicator. The Sleepio algorithm tailors ongoing intervention based on this sleep data and other data about participants' physical and mental health. Sleepio also provides access to online psychoeducation and a clinician-moderated user forum. This intervention has been shown to be as effective as 1-1 CBT-I in the general population. Sleepio has been used in mental health populations but has not yet been tested in people experiencing a first episode of psychosis.

The study aims to use mixed methods to determine how digital CBT-I can be implemented in first episode psychosis services. These data will be integrated to build a logic model, based on the Medical Research Council (MRC) complex interventions framework.

Keyworkers in Esteem FEP services will be approached to identify service users affected by sleep difficulties that may benefit from Sleepio. Service user participants will be recruited through their treatment as usual (TAU) with their Esteem keyworker (sleep monitoring is part of this). Where service users report sleep difficulties, keyworkers will offer an information leaflet about the study and referral into the research study or contact details for researchers (study email address). Keyworkers will record that service users have agreed to keyworkers providing their details to researchers and to being contacted by the researchers in their casefile.

Those service users who wish to find out more about the study and meet eligibility criteria will be sent an easy-read Participant Information Sheet and Consent Form. They will be given the opportunity to ask questions and will be encouraged to speak to others about their potential participation (such as their keyworker). It will be made clear that in consenting to participate they are consenting to participate in sleep assessment, complete symptomatology measures pre- and post-intervention and use the Sleepio intervention. It will be made clear that participation does not affect their TAU. They will provide written consent if they wish to participate. Consenting service user study participants will receive access to Sleepio. They will register for the intervention with a researcher during the baseline symptomology measures assessment session.

They will be given the option of additionally participating in semi-structured interviews prior to and after using the intervention, to talk about their expectations and experiences of Sleepio. Service user participants will not be randomized to treatment. All service user participants will be provided with access to Sleepio. Research will focus on developing a model for the implementation of this intervention.

Keyworkers will be introduced to and supported in their role in referring service users to the study and monitoring use of Sleepio through presentations, psychosocial supervision, and reflection sessions. Keyworkers will be provided with an easy read information sheet which clarifies their role as clinicians (attending a session to reflect on their caseload and service user suitability for the study and providing suitable service users with information about the study) and potentially as research participants (in semi-structured interviews) via email and letter. They will be given the opportunity to ask questions and will be encouraged to speak to others about their potential interview participation (such as their colleagues). They will provide written consent if they wish to participate in semi-structured interviews, to talk about their expectations and experiences of Sleepio use in Esteem.

Primary outcomes comprise implementation data and qualitative data concerning the perspectives of clinicians and service users, which inform the resulting logic model. Secondary outcome data comprises insomnia severity (Insomnia Severity Index), mental health symptomatology (Depression Anxiety and Stress Scales; The Revised Green et al., Paranoid Thoughts Scale (R-GPTS); Specific Psychotic Experiences Questionnaire (SPEQ) - Hallucinations Subscale) and worry about Covid19 (Fear of Covid19 Scale).

ELIGIBILITY:
Inclusion Criteria:

* Service users under the care of Esteem First Episode Psychosis Service in NHS GGC
* Potentially affected by Insomnia Disorder (defined by Sleep Condition Indicator-02 score ≤2)
* Who have access to a device they can use Sleepio on (a computer device with Safari or Google Chrome browser, or an iPhone device).

Exclusion Criteria:

* Moderate to severe learning disability
* Acute Psychosis (recent crisis contact or hospitalisation)
* Incapacity to provide informed consent
* Insufficient English to access intervention
* Organic impairment
* No access to a device which can be used for Sleepio intervention.

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Estimated)
Dates: Start 2021-04-20 (Actual); Primary Completion 2022-04-20 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Implementation data - rates of consenting | Across study timeline (8 months), across 10 weeks for Sleepio specific measures
  Rates of consenting and nonconsenting interested participants
Implementation data - eligibility | 8 months
  Number of eligible vs. ineligible participants and reasons for ineligibility
Implementation data - completion of measures | 8 months
  Participant completion of measures assessment appointments and measures (ISI measure of insomnia severity, DASS-21 measure of mental wellbeing, R-GPTS measure of paranoia, SPEQ measure of hallucination, and Fear of Covid19). This outcome records whether or not these were completed by participants, whereas secondary outcomes 6-10 examine participant scores on these measures.
Implementation data - completion of intervention sessions | Across 10 weeks per participant
  Measures attrition from intervention by recording how many sessions of intervention were completed by participant.
Qualitative data | Across study timeline (8 months), across 12 weeks for service users (pre and post intervention)
  Service user and clinician expectations and experiences of digital CBT-I intervention

SECONDARY OUTCOMES:
Insomnia severity | 10 weeks
  As measured by the Insomnia Severity Index (ISI). Possible scores range from 0 to 28 and higher scores indicate more severe insomnia.
Mental Wellbeing | 10 weeks
  As measured by the Depression, Anxiety and Stress Scales (DASS-21). Possible scores range from 0 to 126 and higher scores indicate more psychological distress. The maximum score on each subscale (depression, anxiety, stress) is 42.
Paranoia symptomatology | 10 weeks
  As measured by the Revised Green et al., Paranoid Thoughts Scale (R-GPTS). Possible scores range from 0 to 72 and higher scores indicate more severe paranoia.
Hallucination symptomatology | 10 weeks
  As measured by the Specific Psychotic Experiences Questionnaire (SPEQ) - Hallucinations subscale. Possible scores range from 0 to 45 and higher scores indicate more severe hallucinatory experience.
Anxiety regarding Covid19 | 10 weeks
  As measured by the Fear of Covid19 Scale. Possible scores range from 7 to 35 and higher scores indicate more fear of Covid19.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Gumley, Principal Investigator — NHS Greater Glasgow and Clyde; University of Glasgow
Locations (2):
- United Kingdom (2):
  - Esteem North, NHS Greater Glasgow and Clyde, Glasgow
  - Esteem South and Clyde, NHS Greater Glasgow and Clyde, Glasgow

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2021-03-12): https://cdn.clinicaltrials.gov/large-docs/01/NCT05050201/Prot_000.pdf